CLINICAL TRIAL: NCT03347786
Title: Intraarterial Verapamil for Neuroprotection in Ischemic Stroke
Brief Title: Verapamil for Neuroprotection in Stroke
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Global Neurosciences Institute (Other)
Responsible Party: Principal Investigator, Mandy Binning, Director, Global Neurosciences Institute, Global Neurosciences Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GNI_verapamil
Record Dates: First submitted 2017-11-09; First posted 2017-11-20 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Each trial participant is randomly assigned to one of two total intervention groups. The first intervention group will receive a dose of 10mg Verapamil, while the second intervention group will receive a dose of 20mg Verapamil. Both treatment groups will have Verapamil administered intra-arterially following mechanical thrombectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Verapamil 10 mg Treatment Group (Experimental): Ischemic stroke patients with large penumbra are offered Verapamil treatment following mechanical thrombectomy. The patient will be randomly assigned an intervention group with the specified dose (10 mg) Verapamil.
  Interventions: Drug: 10 mg Intra-arterial Verapamil
- Verapamil 20 mg Treatment Group (Experimental): Ischemic stroke patients with large penumbra are offered Verapamil treatment following mechanical thrombectomy. The patient will be randomly assigned an intervention group with the specified dose (20 mg) Verapamil.
  Interventions: Drug: 20 mg Intra-arterial Verapamil

INTERVENTIONS:
Drug: 10 mg Intra-arterial Verapamil — Intra-arterial delivery of verapamil following mechanical thrombectomy procedure will be administered at a randomized dose of 10 mg or 20 mg to consenting patients.
  Arms: Verapamil 10 mg Treatment Group
Drug: 20 mg Intra-arterial Verapamil — Intra-arterial delivery of verapamil following mechanical thrombectomy procedure will be administered at a randomized dose of 10 mg or 20 mg to consenting patients.
  Arms: Verapamil 20 mg Treatment Group

SUMMARY:
The purpose of this research study is to test an experimental procedure called intra-arterial delivery of verapamil in patients diagnosed with acute ischemic stroke. This study investigates the safety of intra-arterial delivery of verapamil, a drug used to treat vasospasm (spasm of a blood vessel), and how it affects recovery from stroke. Recruitment is limited to patients that have received mechanical thrombectomy as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* 18 years of age and over
* Acute onset focal neurologic deficit consistent with acute ischemic stroke, or computed tomographic scan consistent with acute cerebral ischemia
* Candidate for mechanical thrombectomy procedure
* Onset of symptoms less than 8 hours
* Measurable neurologic deficit (NIHSS ≥4)
* Willingness to follow up with rehabilitation therapy
* Anticipated life expectancy of at least 3 months

Exclusion Criteria:

* Pregnancy or suspected pregnancy (pregnancy test will be done on women of child-bearing potential)
* Hepatic and/or renal insufficiency (LFT's>3× upper limit of normal; CrCl < 30ml/min)
* Thrombocytopenia (platelet count <75,000/mm3)
* History of intolerance to verapamil
* Previous functional disability (modified Rankin > 1)
* Severe stroke (NIHSS>22)
* Stuporous or comatose
* Unlikely to be available for 90 day follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Bleeding Complications | 3 months
  Bleeding Complications including: symptomatic intracerebral hemorrhage (sICH), and Hemorrhagic Transformation (HT)
Number of Participants with a Serious Adverse Event of Death | 3 months
  Death

SECONDARY OUTCOMES:
Functional Outcomes | 30-days and 90-days
  Change in modified Rankin Scale (mRS) Score
Functional Outcomes | 30-days and 90-days
  Change in National Institutes of Health Stroke Scale (NIHSS) Score
Neuroimaging | 180 Days, 365 Days
  MRI/ CT Scan

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - AtlantiCare Regional Medical Center, Atlantic City, New Jersey
  - St Mary Medical Center, Langhorne, Pennsylvania
  - Crozer Chester Medical Center, Upland, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared as this is a pilot study.